CLINICAL TRIAL: NCT03001661
Title: A Randomised Controlled Trial of a Synthetic Osmotic Cervical Dilator for Induction of Labour in Comparison to Dinoprostone Vaginal insErt: the SOLVE Trial
Brief Title: An RCT of a Synthetic Osmotic Cervical Dilator for Induction of Labour in Comparison to Dinoprostone Vaginal insErt
Acronym: SOLVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Collaborators: University of Birmingham (Other); Medicem International CR s.r.o. (Industry)
Responsible Party: Principal Investigator, Professor Janesh Gupta, Professor of Obstetrics and Gynaecology, Birmingham Women's and Children's NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Solve
Record Dates: First submitted 2016-11-11; First posted 2016-12-23 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Induction of Labor Affected Fetus / Newborn
Keywords: Propess; Dilapan-S; Dinoprostone; Labour; Induction; Child birth
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propess (Active Comparator): Control intervention: Propess® (dinoprostone) Slow release vaginal drug delivery system (Prostaglandin E2).
  Interventions: Drug: Dinoprostone
- Dilapan-S (Experimental): Experimental intervention: DILAPAN-S® A synthetic osmotic cervical dilator for insertion into the cervical canal, using as many rods as necessary.
  Interventions: Device: Dilapan-S

INTERVENTIONS:
Device: Dilapan-S — DILAPAN-S® is a non-pharmacological synthetic rod, which is inserted into the cervical canal and through the internal os, for cervical ripening prior to induction. Its mode of action consists in the hydrophilic properties of the device absorbing fluids from surrounding tissue structures, thus expanding the volume of DILAPAN-S® sticks, usually within a 12-hour period. Subsequently it exerts radial pressure on the surrounding structures (cervix) to dilate progressively. Endocervical pressure on the cervix results not only in its mechanical dilatation but the pressure on the endocervical structures also stimulates the production of endogenous PGs and promotes cervical ripening through its collagenolytic action.
  Other Names: Synthetic Osmotic Cervical Dilator
  Arms: Dilapan-S
Drug: Dinoprostone — Dinoprostone slow release 10mg vaginal insert is currently the standard method used for induction of labour in the NHS, particularly in nulliparous woman.
  Other Names: Propess
  Arms: Propess

SUMMARY:
Induction of labour (where labour is started artificially) is traditionally carried out with a range of different drugs or by surgery (rupturing the membranes or 'waters'). Dilapan-S is a mechanical device, known as an osmotic cervical dilator, which provides an alternative to drugs or surgery. Thin rods of an absorbent material (no active drug present) are inserted into the neck of the womb (cervix) and, as they absorb fluid, they swell and mimic the natural process of 'ripening' (or preparing) the cervix. This initial process is important before contractions begin. Unlike drugs, Dilapan-S does not cause premature contractions that, when too frequent, may cause the baby to become distressed. The project will compare cervical ripening using Dilapan-S with the standard use prostaglandin drug. Women with a single pregnancy, who require induction of labour, and who are not considered high risk, will be invited to participate. Investigators hope to recruit 860 women from UK maternity units over 2 years. Participants will have an equal chance of being randomised to the drug, which is standard practice, or the cervical dilator. The speed in which labour commences, the mode of delivery and any side effects will be compared. Importantly, investigators shall also assess patient satisfaction and anxiety during the induction process, by asking participants to complete a short questionnaire about their experience before they go home after having their baby. If osmotic dilators are effective investigators expect NICE to consider them an option alongside other cervical ripening methods.

DETAILED DESCRIPTION:
Prospective, Phase III, UK, Open, Multicentre, Superiority, Randomised Controlled Trial of a CE marked medical device and an Investigational Medicinal Product (CTIMP).

Potentially eligible patients will be identified by their obstetrician or midwife, based on the need for induction of labour. Once the decision to induce labour is made, women will be approached to participate in the trial and will be given a patient information leaflet (PIL) enclosed in the induction admission letter. Patients wishing to enter the trial will be confirmed for eligibility by an obstetrician. Prior to patients undertaking any trial-related procedures, informed consent will be obtained.

Participants will then be randomised in a 1:1 ratio to either 1) synthetic osmotic cervical dilator or 2) a 10-mg controlled-release dinoprostone vaginal insert. Randomisation will be provided by a computer generated programme. A research assistant discloses the nature of the assignment only after enrolment. Investigators have calculated that 860 patients (430 in each arm) will need to be recruited over a 2 year period. Given the nature of the intervention, the SOLVE trial will not be a blinded trial.

Full data collection will be conducted for those patients giving informed consent, from medical records. This will include baseline data, and details of mother and child at birth. Patients will also be asked to complete a maternal satisfaction questionnaire before they are discharged. There will be no further follow-up of patients post-discharge from care unless a Serious Adverse Event requires this. If the patient withdraws her consent during the study, data collection will be stopped. Only anonymised data will be entered into the Case Report Forms (CRFs) by the study team. Details of all patients approached about the trial will be recorded on the trial Screening Log, and fully anonymised copies returned to the trials office for review.

ELIGIBILITY:
Inclusion criteria

Women must meet the following criteria prior to initiation of IoL:

1. ≥ 16 years of age
2. Able to provide informed consent
3. Singleton pregnancy
4. Indication for IoL
5. Pregnancy ≥ 37.0 weeks (assessed as an agreed gestational age by ultrasound dating scan)
6. Living fetus with vertex presentation
7. Intact membranes

Exclusion criteria

1. Women already receiving oxytocin
2. Diagnosis of fulminant preeclampsia / eclampsia
3. Contraindication to DINOPROSTONE or DILAPAN
4. If DINOPROSTONE for IoL is non-compliant with local policy
5. Enrolled in other randomised controlled trials of an IMP or device for cervical ripening or induction of labour

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Failure to achieve vaginal delivery | 1 year from study completion
  To evaluate the efficacy of the use of the synthetic osmotic cervical dilator in cervical ripening, prior to induction of labour, in comparison to dinoprostone vaginal insert in the parameter of failure to achieve vaginal delivery

SECONDARY OUTCOMES:
Failure to achieve vaginal delivery within 24, 36 and 48 hours from randomisation | 24, 36 and 48 hours
  Failure to achieve vaginal delivery within 24, 36 and 48 hours from randomisation
caesarean section | 24 and 64 hours
  caesarean section undertaken between randomisation and delivery of fetus. The maximum time period for use of trial induction methods is 64 hours for Propess and 24 for Dilapan-S, thus C-section should typically have taken place by these time periods.
instrumental delivery | 24 and 64 hours
  instrumental delivery undertaken between randomisation and delivery of fetus. The maximum time period for use of trial induction methods is 64 hours for Propess and 24 for Dilapan-S, thus instrumental delivery should typically have taken place by these time periods.
spontaneous delivery | 0 - 64 hours
  spontaneous delivery between randomisation and delivery of fetus. The maximum time period for use of intervention is 64 hours, so spontaneous labour should have taken place by this stage.
Change in Bishop Score | 0 hours, 12 hours, 24 hours, 32 hours, 56 hours, 64 hours.
  change in Bishop Score compared at initiation of cervical ripening (i.e. randomisation) and completion of cervical ripening (i.e. when treatment is completed at 12 or 24 hours with Dilapan-S, or at 24, 32, 56 or 64 hours with Propess; or once labour is initiated - whichever comes first)
Total duration of intervention received | 0 hours, 12 hours, 24 hours, 32 hours, 56 hours, 64 hours.
  Total duration of intervention received (i.e. randomisation) and completion of cervical ripening (i.e. when treatment is completed at 12 or 24 hours with Dilapan-S, or at 24, 32, 56 or 64 hours with Propess; or once labour is initiated - whichever comes first)
Use of Oxytocin | 0 hours, 12 hours, 24 hours, 32 hours, 56 hours, 64 hours.
  Use of Oxytocin for induction and/or augmentation of labour from randomisation to completion of induction (i.e. when treatment is completed at 12 or 24 hours with Dilapan-S, or at 24, 32, 56 or 64 hours with Propess; or once labour is initiated - whichever comes first)
Use of Analgesia | 0 - 64 hours approx.
  Use of Analgesia during induction and/or labour (from randomisation until delivery of fetus).
Amniotomy undertaken | 0 hours, 12 hours, 24 hours, 32 hours, 56 hours, 64 hours.
  Amniotomy undertaken for induction and/or augmentation of labour from randomisation to completion of induction (i.e. when treatment is completed at 12 or 24 hours with Dilapan-S, or at 24, 32, 56 or 64 hours with Propess; or once labour is initiated - whichever comes first)
maternal and neonatal safety: SAEs recorded from randomisation up to discharge, and resolution of SAE. | 0 hours up to discharge (typically 4 days for c-section) or resolution of SAE (approx 2 weeks).
  maternal and neonatal safety: SAEs recorded from randomisation up to discharge, and resolution of SAE.
maternal satisfaction with cervical ripening | 1hr to 4 days
  maternal satisfaction with cervical ripening collected after delivery, prior to discharge.
fetal status after delivery | recorded on delivery of fetus
  fetal status after delivery recorded on delivery of fetus

CONTACTS AND LOCATIONS:
Overall Officials: Janesh Gupta, MD, Principal Investigator — Birmingham Women's and Children's Hospital NHS Foundation Trust
Locations (1):
- Birmingham Women's and Children's NHS Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Investigators will not be sharing individual patient data with other research studies

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264

DOCUMENTS (2):
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT03001661/Prot_000.pdf
  • Informed Consent Form (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT03001661/ICF_001.pdf